CLINICAL TRIAL: NCT02153125
Title: Eplerenone For the Treatment of Chronic Central Serous Chorioretinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michaella Goldstein, Deputy Head Department of Ophthalmology, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0405-13-TLV
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Eplerenone (Experimental): 25mg eplerenone given daily for a week, followed by 50mg given for a total of 3 months since commencement of treatment
  Interventions: Drug: Eplerenone
- Placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Eplerenone
  Arms: Eplerenone

SUMMARY:
The aim of the study is to determine the efficacy and safety in treating patients with chronic central serous chorioretinopathy with the drug eplerenone.

DETAILED DESCRIPTION:
* The goal of the study is to examine the short-term effects and safety of eplerenone, a systemic anti-aldosterone medication, in a group of patients with central serous chorioretinopathy (CSCR).
* There is currently no standard treatment or therapy for chronic CSCR, a potentially debilitating eye disease.
* There is evidence that high blood serum corticosteroid levels can cause or worsen CSCR
* Eplerenone, a mineralocorticoid receptor antagonist, has been shown to be of visual and anatomic benefit in a small series of 4 patients with chronic CSCR, suggesting that decreasing mineralocorticoid action in the eye may improve signs and symptoms of CSCR
* The study's aim is to evaluate a standardized dose of eplerenone in a controlled prospective fashion for chronic CSCR.
* The study consists of taking a standard dose of eplerenone, 25mg once daily for a week, followed by 50mg once daily, for a total of 3 months
* Patients will be monitored for efficacy and side effects from the beginning of treatment and for 6 months

ELIGIBILITY:
Inclusion Criteria:

* Chronic central serous chorioretinopathy (CSCR): Previous diagnosis of CSCR, persistent subretinal fluid on OCT for more than 4 months after initial presentation to the eye clinic

Exclusion Criteria:

* Other retinal disease
* Choroidal neovascularization
* Diabetes
* A history of uveitis
* Ocular surgery in the prior 3 months
* Allergy to fluorescein or indocyanine green
* Pregnancy, lactation or female patients in fertility age not treated with contraceptive pills
* Creatinine clearance < 50 ml/min
* Hyperkalemia > 5 mmol/l
* Patients treated with drugs deactivated by cytochrome P450 3A4 (CYP3A4)
* Serum creatinine > 2 mg/dl in men or > 1.8 mg/dl in women
* Treatment with potassium sparing agents or potassium
* Treatment with Angiotensin converting enzyme (ACE)/angiotensin II receptor blocker (ARB) inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Decrease of at least 10% in subretinal fluid thickness as measured by optical coherence tomography (OCT) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Souraski Medical Center, Tel Aviv, Israel, Israel

REFERENCES:
- [Background] Zhao M, Celerier I, Bousquet E, Jeanny JC, Jonet L, Savoldelli M, Offret O, Curan A, Farman N, Jaisser F, Behar-Cohen F. Mineralocorticoid receptor is involved in rat and human ocular chorioretinopathy. J Clin Invest. 2012 Jul;122(7):2672-9. doi: 10.1172/JCI61427. Epub 2012 Jun 11. PMID 22684104
- [Background] Gemenetzi M, De Salvo G, Lotery AJ. Central serous chorioretinopathy: an update on pathogenesis and treatment. Eye (Lond). 2010 Dec;24(12):1743-56. doi: 10.1038/eye.2010.130. Epub 2010 Oct 8. PMID 20930852
- [Background] Chan WM, Lai TY, Lai RY, Liu DT, Lam DS. Half-dose verteporfin photodynamic therapy for acute central serous chorioretinopathy: one-year results of a randomized controlled trial. Ophthalmology. 2008 Oct;115(10):1756-65. doi: 10.1016/j.ophtha.2008.04.014. Epub 2008 Jun 5. PMID 18538401
- [Background] Reibaldi M, Cardascia N, Longo A, Furino C, Avitabile T, Faro S, Sanfilippo M, Russo A, Uva MG, Munno F, Cannemi V, Zagari M, Boscia F. Standard-fluence versus low-fluence photodynamic therapy in chronic central serous chorioretinopathy: a nonrandomized clinical trial. Am J Ophthalmol. 2010 Feb;149(2):307-315.e2. doi: 10.1016/j.ajo.2009.08.026. Epub 2009 Nov 6. PMID 19896635
- [Background] Robertson DM, Ilstrup D. Direct, indirect, and sham laser photocoagulation in the management of central serous chorioretinopathy. Am J Ophthalmol. 1983 Apr;95(4):457-66. doi: 10.1016/0002-9394(83)90265-9. PMID 6682293
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203